CLINICAL TRIAL: NCT00005756
Title: Epidemiology of Coronary Calcification in the Elderly
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anne B. Newman, Professor of Epidemiology, University of Pittsburgh
Other Study IDs: 5111; R01HL064587 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Arteriosclerosis; Coronary Disease; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Coronary Disease; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the prevalence and prognostic value of subclinical atherosclerosis in the Pittsburgh SHEP cohort and a cohort of normal controls.

DETAILED DESCRIPTION:
BACKGROUND:

This is an ancillary study to the Systolic Hypertension in the Elderly Program (SHEP)

DESIGN NARRATIVE:

Continued annual telephone follow-up of the remaining 178 Pittsburgh SHEP participants and 168 controls will be conducted . A final clinic visit will include measures of coronary and aortic calcification using electron beam computed tomography (CT), pulse wave velocity as a measure of aortic stiffening and cognitive function testing. For the Pittsburgh SHEP cohort, the antihypertensive treatment effect has been striking with event rates for the active and placebo groups continuing to diverge beyong the end of SHEP. Successful demonstration of a treatment effect on coronary calcium scores would be the first randomized data showing an antihypertensive effect directly in the coronary arteries. Risk factors for coronary calcification will be evaluated, producing data of a type not yet available in the literature for older adults and not being collected in any other ongoing studies of the elderly. The added measures of vascular stiffness will supplement the extensive data on subclinical atherosclerosis already available for this cohort. The extent to which these measures predict cardiovascular events will be evaluated. The study has been renewed through July 2006.

Since hypertension and aging are associated with cognitive impairment and vascular dementia, SHEP participants assigned to the placebo group are expected to have lower cognitive function compared to those assigned to active treatment. Among both hypertensive and normotensive groups, lower cognitive function among those with evidence of subclinical atherosclerosis is expected.

Finally, members of the cohort who were originally normotensive at study entry are now developing systolic hypertension. These subjects will allow a prospective evaluation of risk factors for systolic hypertension. Continued study of this cohort into their 80s will provide unique data on the risks and etiology of systolic hypertension, the efficacy of its treatment and the prognostic value of a number of measures of subclinical atherosclerosis. It is predicted that the results will be directly applicable to the largest growing segment of the U.S. population.

ELIGIBILITY:
Participating in the Cardiovascular Health Study (CHS) at the University of Pittsburgh Site.

Inclusion criteria:

Age 65 or older in 1989-90 Able to give informed consent Able to travel to study site No plans to move from the area within 3 years of CHS enrollment

Exclusion criteria:

Inability to give informed consent at time of EBCT scan Unable to travel to study center Lives in nursing home.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 614 older adults aged, on average, 80 years (range, 67 to 99 years); 367 (60%) were women, and 143 (23%) were black.
Sampling Method: Non-Probability Sample
Dates: Start 1999-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne B. Newman, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Newman AB, Naydeck BL, Sutton-Tyrrell K, Feldman A, Edmundowicz D, Kuller LH. Coronary artery calcification in older adults to age 99: prevalence and risk factors. Circulation. 2001 Nov 27;104(22):2679-84. doi: 10.1161/hc4601.099464. PMID 11723018
- [Background] Newman AB, Naydeck BL, Sutton-Tyrrell K, Edmundowicz D, O'Leary D, Kronmal R, Burke GL, Kuller LH. Relationship between coronary artery calcification and other measures of subclinical cardiovascular disease in older adults. Arterioscler Thromb Vasc Biol. 2002 Oct 1;22(10):1674-9. doi: 10.1161/01.atv.0000033540.89672.24. PMID 12377748
- [Background] Newman AB, Naydeck BL, Whittle J, Sutton-Tyrrell K, Edmundowicz D, Kuller LH. Racial differences in coronary artery calcification in older adults. Arterioscler Thromb Vasc Biol. 2002 Mar 1;22(3):424-30. doi: 10.1161/hq0302.105357. PMID 11884285
- [Background] Rosano C, Aizenstein HJ, Cochran JL, Saxton JA, De Kosky ST, Newman AB, Kuller LH, Lopez OL, Carter CS. Event-related functional magnetic resonance imaging investigation of executive control in very old individuals with mild cognitive impairment. Biol Psychiatry. 2005 Apr 1;57(7):761-7. doi: 10.1016/j.biopsych.2004.12.031. PMID 15820233
- [Background] Rosano C, Aizenstein H, Cochran J, Saxton J, De Kosky S, Newman AB, Kuller LH, Lopez OL, Carter CS. Functional neuroimaging indicators of successful executive control in the oldest old. Neuroimage. 2005 Dec;28(4):881-9. doi: 10.1016/j.neuroimage.2005.05.059. Epub 2005 Oct 12. PMID 16226041